CLINICAL TRIAL: NCT06387355
Title: Diagnosis and Treatment of Coronary Artery Disease in Severe Peripheral Artery Disease After Lower Extremity Revascularization
Brief Title: Diagnosis and Treatment of CAD in Severe PAD After Lower Extremity Revascularization
Acronym: CAD in sPAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Intent to fund was rescinded
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-006-23S
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Artery Disease; Coronary Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease | interventions — Angiography

STUDY DESIGN:
Intervention Model Description: This will be a parallel interventional model to assign participants to a treatment strategy in a clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Treatment Strategy (Experimental): This arm will have a coronary CTA with FFR-CT with selective coronary artery revascularization plus optimal medical therapy after lower extremity revascularization
  Interventions: Diagnostic Test: Coronary computed topography (CT) angiography with FFR-CT
- Standard (No Intervention): This arm will have optimal medical therapy after lower extremity revascularization

INTERVENTIONS:
Diagnostic Test: Coronary computed topography (CT) angiography with FFR-CT — The investigational treatment strategy will have a coronary CT angiography diagnostic imaging with computational analysis FFR-CT (Fractional Flow Reserve from the coronary CTA)
  Arms: Investigational Treatment Strategy

SUMMARY:
Peripheral artery disease, lack or blood flow to the legs, has a high prevalence in the Veteran population. In patients with severe peripheral artery disease that requires an endovascular or surgical intervention for lower leg revascularization, the long-term mortality of approximately 50% is worse that most cancers. The goal of this study is to develop a management strategy to improve cardiovascular outcomes in this high-risk peripheral artery disease population after lower extremity revascularization.

DETAILED DESCRIPTION:
This study will be to conduct a randomized, controlled, multi-center clinical trial to evaluate a non-invasive management strategy of a computed topography (CT) scan of the coronary arteries and computational analysis of coronary perfusion with selective coronary revascularization plus optimal medical therapy compared to optimal medical therapy. Therefore, this study will provide the opportunity for Veterans to participate in a clinical trial to reduce the very high cardiac-related mortality rate in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 50 to 85
* Severe intermittent claudication with ABI < 0.6 or monophasic waveform if non-compressible and TBI < 0.6
* Chronic limb threatening ischemia (CLTI) with pain at rest (Rutherford Category 4) with ABI < 0.5 or TBI < 0.6
* CLTI with minor tissue loss (Rutherford Category 5) with ABI < 0.5 or TBI < 0.6
* Completed Lower Extremity Revascularization and enrolled within 45 days
* The patient or legal representative will provide informed written consent
* The patient has a life expectancy of at least 1 year

Exclusion Criteria:

* Major tissue loss of the ischemic limb (Rutherford Category 6)
* Uncompensated congestive heart failure (NYHA class IV)
* Myocardial infarction or stroke within the past 90 days
* Prior coronary artery bypass graft (CABG) revascularization surgery
* Prior percutaneous coronary intervention (PCI) with angioplasty or stenting
* Presence of a pacemaker
* Congestive heart failure with Ejection Fraction < 30%
* Elevated liver function tests more than twice the upper limit of normal
* Severe Chronic renal disease (Glomerular Filtration Rate, GFR < 30) or on hemodialysis
* Pregnancy, Human Immunodeficiency Virus, or organ transplant recipients
* Current malignancy or malignancy within the last two years unless the treating oncologic physician provides prognosis of an anticipated 2- year survival (i.e., adequately treated non-melanoma skin cancer or adequately treated prostate cancer without metastatic disease)
* Any condition the review panel determines would make the patient unsuitable for participation in the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 2 years
  cardiovascular-related death or myocardial infarction

SECONDARY OUTCOMES:
Cardiovascular-related death | 2 years
  death related to cardiovascular disease (i.e., heart attack)
Myocardioal infarction | 2 years
  heart attack
All-cause mortality | 2 years
  death related to any cause
Amputation-free survival | 2 years
  freedom from major amputation

CONTACTS AND LOCATIONS:
Overall Officials: Clay Quint, MD PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (7):
- United States (7):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
The overall data will be shared and reported, but not individual participant data.